CLINICAL TRIAL: NCT05896163
Title: A PHASE 1b/2, OPEN-LABEL STUDY OF PF-07901801 IN COMBINATION WITH GLOFITAMAB AFTER A FIXED, SINGLE DOSE OF OBINUTUZUMAB IN PARTICIPANTS WITH RELAPSED/REFRACTORY DIFFUSE LARGE B CELL LYMPHOMA NOT ELIGIBLE FOR STEM CELL TRANSPLANTATION
Brief Title: A Study to Learn About the Effects of Two Study Medicines (Maplirpacept [PF-07901801] And Glofitamab) When Given Together In People With Relapsed Or Refractory Diffuse Large B Cell Lymphoma.
Acronym: MAPtivate-6
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4971006; 2022-502822-41-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-05-10; First posted 2023-06-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: DLBCL; Lymphoma; Relapsed; Refractory; CD20; CD3; CD47; Glofitamab; Obinutuzumab; Maplirpacept
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Recurrence | interventions — glofitamab; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Open label/randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b (Experimental): Participants will be allocated to sequential dose levels of PF-07901801, administered in combination with fixed doses of glofitamab after a dose of obinutuzumab, to select doses of PF-07901801 for further evaluation in Phase 2. Approximately 20 participants will be enrolled.
  Interventions: Drug: maplirpacept (PF-07901801); Drug: Glofitamab; Drug: Obinutuzumab
- Phase 2 (Experimental): Participants will be randomized to 1 of 3 different dose levels of PF-07901801 which will be administered in combination with fixed doses of glofitamab after a dose of obinutuzumab. Approximately 50 participants will be enrolled.
  Interventions: Drug: maplirpacept (PF-07901801); Drug: Glofitamab; Drug: Obinutuzumab

INTERVENTIONS:
Drug: maplirpacept (PF-07901801) — Intravenous infusion
Drug: Glofitamab — Intravenous infusion
  Other Names: Columvi
Drug: Obinutuzumab — Intravenous infusion
  Other Names: Gazyva

SUMMARY:
The purpose of this study is to learn about the effects of two study medicines (maplirpacept [PF-07901801] and glofitamab) when given together for the treatment of diffuse large B-cell lymphoma (DLBCL) that is relapsed or is refractory. Relapsed means has returned after last treatment. Refractory means that it has not responded to last treatment. The two study medicines are given after a single dose of obinutuzumab which is the third study medicine.

DLBCL is a type of non-Hodgkin lymphoma (NHL). NHL is a cancer of the lymphatic system. It develops when the body makes abnormal B lymphocytes. These lymphocytes are a type of white blood cell that normally help to fight infections.

This study is seeking adult participants who:

* Have histologically confirmed diagnosis of DLBCL
* Have received at least two first lines of treatment for NHL.
* Are unable or unwilling to undergo a stem cell transplant or CAR-T cell therapy.

Stem cell transplant is a procedure in which a patient receives healthy blood-forming cells to replace their own stem cells that have been destroyed by treatment.

A CAR-T therapy is a type of treatment in which a patient's T cells are changed in the laboratory so they will attack cancer cells.

Everyone in this study will receive all three medicines at the study site by intravenous (IV) infusion which is given directly into a vein. The two study medicines (maplirpacept [PF-07901801] and glofitamab) will be given in 21-day cycles.

At Cycle 0, participants will receive a single dose of obinutuzumab pre-treatment followed by two step-up doses of glofitamab. The combination of maplirpacept (PF-07901801) with glofitamab full dose will be administered for the first time at Cycle 1 Day 1.

Maplirpacept (PF-07901801) will be given weekly for the first three cycles and then every three weeks. Glofitamab will be given every 3 weeks for approximately 9 months. Thereafter participants will continue to receive maplirpacept alone.

Maplirpacept (PF-07901801) will be given at different doses to different participants. Everyone taking part will receive the same fixed doses of glofitamab and obinutuzumab studied in patients with DLBCL.

The study will compare the experiences of people receiving different doses of maplirpacept (PF-07901801). This will help to determine what dose is safe and effective when given with the other 2 study medicines.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase 1b/2 study to evaluate the safety, tolerability and potential clinical benefits of maplirpacept PF-07901801, an anti-CD47 molecule, in combination with fixed doses of glofitamab after a single dose of obinutuzumab in participants with relapsed/refractory (R/R) DLBCL not eligible for or unwilling to undergo high dose chemotherapy and subsequent autologous stem cell transplantation (ASCT) or unable to receive approved chimeric antigen receptor T-cell (CAR-T) therapy (for example, due to logistical limitations).

For Phase 1b, participants must have previously received at least 2 prior systemic treatment regimen. For Phase 2, participants must have received at least 2 but no more than 4 prior systemic treatment regimens. All participants must have previously received an anti-CD20 containing regimen.

Phase 1b will assess dose-limiting toxicities of PF-07901801 when administered in combination with glofitamab, to select doses for the Phase 2 part of the study. Phase 2 will evaluate safety and efficacy to determine the recommended Phase 3 dose of PF-07901801 to be administered in combination with glofitamab.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of DLBCL
* Relapsed or refractory disease
* Participant is not be a candidate for or is unwilling to undergo high dose chemotherapy and subsequent stem cell transplant and/or is unable to receive chimeric antigen receptor (CAR) T-cell therapy
* Previous treatment with at least two prior lines of systemic therapy (for phase 2, at least 2 and no more than 4 prior lines of systemic therapy). Prior therapy must include an anti-CD20 antibody.
* Adequate bone marrow, hepatic and renal function
* Eastern Cooperative Oncology Group (ECOG) ≤2

Key Exclusion Criteria:

* Prior treatment with anti-CD47 and/or prior glofitamab or anti-CD20 x CD3 containing regimen. Refractoriness to an obinutuzumab monotherapy containing regimen.
* Prior allogeneic stem cell transplantation or autologous stem cell transplantation within 12 weeks prior to enrolment
* High Grade B-Cell Lymphoma
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: Number of participants with Dose limiting toxicities (DLT) | 21 days following first PF-07901801 dose
  DLTs are a predefined set of adverse events that are at least possibly related to any or all of the investigational agents.
Phase 2: Objective Response (OR) | Time from the date of first dose of study intervention until the first documentation of disease progression, death, or start of new anticancer therapy (assessed up to approximately 24 months)
  OR defined as proportion of participants with objective response based assessment of complete response (CR) or partial response (PR) according to Lugano Response Classification Criteria 2014.

SECONDARY OUTCOMES:
Phase 1b and Phase 2: Frequency of adverse events (AE) | Time from the date of first dose of study intervention through 28 days after last dose of PF-07901801 or 90 days after last dose of glofitamab or obinutuzumab (assessed up to approximately 24 months)
  Type and severity (severity according to the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], version 5.0). Severity of Cytokine Release Syndrome (CRS) and Immune effector cell-associated neurotoxicity syndrome (ICANS) assessed according to ASTCT criteria.
Phase 1b and Phase 2: Frequency of clinical laboratory abnormalities | Time from the date of first dose of study intervention through 28 days after last dose of PF-07901801 or 90 days after last dose of glofitamab or obinutuzumab (assessed up to approximately 24 months)
  Type and severity (severity according to the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], version 5.0).
Phase 1b: Objective Response (OR) | Time from the date of first dose of study intervention until the first documentation of disease progression, death, or start of new anticancer therapy (assessed up to approximately 24 months)
  OR defined as proportion of participants with objective response based assessment of complete response (CR) or partial response (PR) according to Lugano Response Classification Criteria 2014.
Phase 1b and Phase 2: Duration of Response (DoR) | Time from the date of first dose of study intervention until the first documentation of disease progression, death, or start of new anticancer therapy (assessed up to approximately 24 months)
  DoR defined as the time from the first documentation of OR until progressive disease (PD), or death due to any cause, whichever occurs first.
Phase 1b and Phase 2: Complete Response (CR) | Time from the date of first dose of study intervention until the first documentation of disease progression, death, or start of new anticancer therapy (assessed up to approximately 24 months)
  CR defined per Lugano Response Classification Criteria 2014
Phase 1b and Phase 2: Duration of Complete Response (DoCR) | Time from the date of first dose of study intervention until PD, or death due to any cause, whichever occurs first (assessed up to approximately 24 months)
  DoCR defined as the time from the first documentation of a CR until PD, or death due to any cause, whichever occurs first.
Phase 1b and Phase 2: Progression Free Survival (PFS) | Time from the date of first dose of study intervention until PD, or death due to any cause, whichever occurs first (assessed up to approximately 24 months)
  PFS is defined as the time from the date of first dose until PD per Lugano Response Classification Criteria 2014, or death due to any cause, whichever occurs first.
Phase 1b and Phase 2: Serum Concentration Versus Time Summary of PF-07901801 | Pre and post-infusion on Day 1 of Cycle 1 and 2 (each cycle is 21 days), Pre-infusion on Day 8 of Cycle 1, Pre-infusion on Day 1 of Cycles 3, 4, 5, 7, 10, 13 and every 6 cycle thereafter until end of treatment (approximately 24 months)
  Pre- and post-dose concentrations of PF-07901801
Phase 1b and Phase 2: Number of participants with Anti-Drug Antibody (ADA) against PF-07901801 | On the first day of every 21-day cycle through 5 cycles, then every third cycle from cycle 7 through cycle 13 and then every sixth cycle thereafter until end of PF-07901801 treatment (assessed up to approximately 24 months)
  To evaluate immunogenicity of PF-07901801
Phase 1b and Phase 2: Number of participants with Neutralizing antibody (NAb) for PF-07901801 | On the first day of every 21-day cycle through 5 cycles, then every third cycle from cycle 7 through cycle 13 and then every sixth cycle thereafter until end of PF-07901801 treatment (assessed up to approximately 24 months)
  To evaluate immunogenicity of PF-07901801

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (9):
  - The University of Kansas Hospital, Kansas City, Kansas
  - University of Kansas Hospital Cambridge North Tower A, Kansas City, Kansas
  - Allina Health Cancer Institute - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Siteman Cancer Center, St Louis, Missouri
  - Barnes-Jewish Hospital Parkview Tower, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Princess Alexandra Hospital, Brisbane, Queensland, Australia
- Israel (4):
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB
- Japan (3):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4971006